CLINICAL TRIAL: NCT04890496
Title: Analysis of Hospitalization Data in Zhongshan Ophthalmology Center
Brief Title: Analysis of Hospitalization Data From ZOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: HBD2021
Record Dates: First submitted 2021-03-18; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Ophthalmology; Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- inpatients of ZOC: Patients have retrospective hopitalization record of ZOC from 1998 to 2020.

SUMMARY:
The real-world electronic health records (EHR) were derived from the hospitalization of Zhongshan Ophthalmic Center (ZOC) of Sun Yat-sen University from 1998-2020 to investigate the ophthalmology diagnosis and treatment activities.

ELIGIBILITY:
Inclusion Criteria:

* have retrospective inpatient records of ZOC from 1998 to 2020

Exclusion Criteria:

* Demographic data missing
* Diagnosis data missing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients have retrospective inpatient records of ZOC from 1998 to 2020.
Sampling Method: Non-Probability Sample
Enrollment: 560000 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The prevalence of primary diagnosis | baseline
  calculate the prevalence of the primary diagnosis of inpatient visits

SECONDARY OUTCOMES:
The prevalence of secondary diagnosis | baseline
  calculate the prevalence of the secondary diagnosis of inpatient visits
Demographics | baseline
  Demographics of inpatient visits
costs of inpatient visits | baseline
  costs of inpatient visits

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Ph.D, M.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China